CLINICAL TRIAL: NCT01642238
Title: Randomized, Crossover Study of the Antithrombotic Effects of Ticagrelor Plus Aspirin Versus Clopidogrel Plus Aspirin When Administered With Bivalirudin
Brief Title: Antithrombotic Effects of Ticagrelor Versus Clopidogrel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Juan J Badimon (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Juan J Badimon, Director, AtheroThrombosis Research Unit, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GCO 12-0732; ISSBRIL0067
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-06

CONDITIONS: Acute Coronary Syndrome
Keywords: Antiplatelet; ticagrelor; clopidogrel; bivalirudin; thrombosis
MeSH Terms: conditions — Acute Coronary Syndrome; Thrombosis | interventions — Ticagrelor; bivalirudin; Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor + ASA + Bivalirudin (Experimental): Single loading dose of Ticagrelor (180 mg given as two 90 mg tablets), plus single dose of ASA (one 81 mg tablet) + bivalirudin administered as 0.75 mg/kg IV bolus followed by 1.75 mg/kg/hour for 1 hour.
  Interventions: Drug: Ticagrelor + ASA + Bivalirudin
- Clopidogrel + ASA + Bivalirudin (Active Comparator): Single loading dose of Clopidogrel (600 mg given as two 300 mg tablets), plus single dose of ASA (one 81 mg tablet) + bivalirudin administered as 0.75 mg/kg IV bolus followed by 1.75 mg/kg/hour for 1 hour.
  Interventions: Drug: Clopidogrel + ASA + Bivalirudin

INTERVENTIONS:
Drug: Ticagrelor + ASA + Bivalirudin — Single loading dose of Ticagrelor (180 mg given as two 90 mg tablets), plus single dose of ASA (one 81 mg tablet) + bivalirudin administered as 0.75 mg/kg IV bolus followed by 1.75 mg/kg/hour for 1 hour.
  Other Names: Brilinta (ticagrelor; Aspirin (ASA); Angiomax (bivalirudin)
  Arms: Ticagrelor + ASA + Bivalirudin
Drug: Clopidogrel + ASA + Bivalirudin — Single loading dose of Clopidogrel (600 mg given as two 300 mg tablets), plus single dose of ASA (one 81 mg tablet) + bivalirudin administered as 0.75 mg/kg IV bolus followed by 1.75 mg/kg/hour for 1 hour.
  Other Names: Plavix (clopidogrel); Aspirin (ASA); Angiomax (bivalirudin)
  Arms: Clopidogrel + ASA + Bivalirudin

SUMMARY:
The purpose of this study is to determine whether treatment with ticagrelor (plus aspirin and bivalirudin) is more effective than treatment with clopidogrel (plus aspirin and bivalirudin).

DETAILED DESCRIPTION:
The HORIZONS-AMI Trial compared the effectiveness of heparin plus a glycoprotein IIb/IIIa inhibitor (GPI) versus bivalirudin in acute myocardial infarction (AMI) patients undergoing stent deployment 1. Overall the data showed benefits associated with the bivalirudin treatment with lower rates of all-cause mortality, cardiac mortality, re-infarction and non-CABG related major bleeding; However, the data seems to indicate a non-significant increase in acute stent thrombosis in the bivalirudin group. This observation seems to suggest the potential benefits of adding an antiplatelet agent to bivalirudin. A study by Dangas G et al found that in the HORIZONS-AMI patients, the group receiving 600 mg loading-dose of clopidogrel had significantly lower 30-day unadjusted rates of mortality, reinfarction and stent thrombosis than the 300 mg loading-dose group, without increase in bleeding rate. Furthermore, even though the benefits of bivalirudin were independent of the clopidogrel loading dose; the 600mg LD was associated with more benefits with both anticoagulation regimens. Similar observations have been reported in the ARMYDA-6 MI study.

It is our hypothesis that using ticagrelor instead of clopidogrel, given its more potent and faster activity, would have greater antithrombotic activity and therefore may reduce the rate of acute stent thrombosis when administered in combination with bivalirudin + ASA in AMI patients. To investigate this hypothesis, we will compare the antithrombotic effects of ticagrelor with clopidogrel, when administered in combination with ASA and bivalirudin, in healthy human volunteers using a cross-over study design. The antithrombotic activity will be assessed pre-treatment and 2-hours and 24-hours post treatment, using methodologies including Badimon Perfusion chamber, VerifyNow P2Y12 assay, platelet aggregation with Multiplate Analyzer and Thromboelastography.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers between 18 and 65 years old.
* Body mass index (BMI) 18 - 30 kg/m2 inclusive.
* Healthy as assessed by a detailed medical history and physical examination.
* Laboratory est results within the normal range.
* Ability to provide signed informed consent.

Exclusion Criteria:

* History of clinically relevant disease, bleeding, acute infectious disease or signs of acute illness.
* Allergy or hypersensitivity to aspirin or thienopyridines, or atopy diagnosed by a physician.
* Use of medication within one month prior to study drug administration.
* History of drug abuse or alcohol consumption >20 g/day.
* Inability to abstain from intensive muscular effort or sport competition.
* Loss of >400 mL blood or blood donation within 3 months.
* Positive serology for hepatitis B (HBs Ag) or hepatitis C.
* Conditions associated with hemorrhagic risk.
* Positive pregnancy test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Badimon, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Zafar MU, Vorchheimer DA, Tewar MP, Giannarelli C, Crippa M, Sartori S, Rodriguez D, Baber U, Mehran R, Badimon JJ. Ticagrelor reduces thrombus formation more than clopidogrel, even when co-administered with bivalirudin. Thromb Haemost. 2014 Nov;112(5):1069-70. doi: 10.1160/TH14-03-0269. Epub 2014 Aug 7. No abstract available. PMID 25104302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 healthy volunteers recruited between July 2012 and March 2013
Groups:
- Ticagrelor, Then Clopidogrel; Clopidogrel, Then Ticagrelor: Acute antithrombotic effects of ticagrelor (180 mg + 90 mg) versus clopidogrel (600mg), when coadministered with aspirin (81mg) and bivalirudin (weight-adjusted clinical dose, given as bolus plus 1-hour infusion) with a 1-2 week washout period in between.
Period: First Intervention (1 Day)
Arm/Group | Ticagrelor, Then Clopidogrel | Clopidogrel, Then Ticagrelor
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: Washout (1-2 Weeks)
Arm/Group | Ticagrelor, Then Clopidogrel | Clopidogrel, Then Ticagrelor
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Ticagrelor, Then Clopidogrel | Clopidogrel, Then Ticagrelor
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Antithrombotic Effects: Acute antithrombotic effects of ticagrelor (180 mg + 90 mg) versus clopidogrel (600mg), when coadministered with aspirin (81mg) and bivalirudin (weight-adjusted clinical dose, given as bolus plus 1-hour infusion) using a randomized, two-treatment, two-period, cross-over design in healthy volunteers.
Arm/Group | Antithrombotic Effects
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 31.2 [26.8 to 35.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Body mass index [Mean (Full Range); unit: kg/m^2] | 27.0 [24.9 to 29.1]

OUTCOME MEASURES:

1. Primary Outcome: Platelet-thrombus Formation in an ex Vivo Model of Thrombosis
Description: Change in thrombus size at 1 hour as compared to Pre-treatment baseline, where a positive change represents a decrease in thrombus size.
Time Frame: Pre-treatment baseline and 1 hour
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Ticagrelor + ASA + Bivalirudin | Clopidogrel + ASA + Bivalirudin
Number analyzed (Participants) | 15 | 15
percent change | 56.3 [43.5 to 69.0] | 35.2 [23.9 to 46.5]

2. Primary Outcome: Platelet-thrombus Formation in an ex Vivo Model of Thrombosis
Description: Change in thrombus size at 24 hours as compared to Pre-treatment baseline, where a positive change represents a decrease in thrombus size.
Time Frame: Pre-treatment baseline and 24 hrs post treatment
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Ticagrelor + ASA + Bivalirudin | Clopidogrel + ASA + Bivalirudin
Number analyzed (Participants) | 15 | 15
percent change | 34.1 [24.3 to 43.9] | 18.5 [4.2 to 32.7]

3. Secondary Outcome: Platelet Reactivity
Description: Platelet reactivity measured by VerifyNowP2Y12 assay measuring percent inhibition
Time Frame: Pre-treatment baseline
Measure: Number (95% Confidence Interval); unit: percent inhibition
Arm/Group | Ticagrelor + ASA + Bivalirudin | Clopidogrel + ASA + Bivalirudin
Number analyzed (Participants) | 15 | 15
percent inhibition | 2.9 [0.5 to 5.3] | 3.7 [0.9 to 6.6]

4. Secondary Outcome: Platelet Reactivity
Description: Platelet reactivity measured by VerifyNowP2Y12 assay measuring percent inhibition
Time Frame: 1 hr post-treatment
Measure: Mean (95% Confidence Interval); unit: percent inhibition
Arm/Group | Ticagrelor + ASA + Bivalirudin | Clopidogrel + ASA + Bivalirudin
Number analyzed (Participants) | 15 | 15
percent inhibition | 69.4 [52.9 to 85.9] | 20.1 [14.5 to 25.8]

5. Secondary Outcome: Platelet Reactivity
Description: Platelet reactivity measured by VerifyNowP2Y12 assay measuring percent inhibition
Time Frame: 24-hours post-treatment
Measure: Mean (95% Confidence Interval); unit: percent inhibition
Arm/Group | Ticagrelor + ASA + Bivalirudin | Clopidogrel + ASA + Bivalirudin
Number analyzed (Participants) | 15 | 15
percent inhibition | 67.4 [54.7 to 80.1] | 53.4 [38.7 to 68.1]

6. Secondary Outcome: Blood Thrombogenicity
Description: Coagulation times, assessed using the ROTEM thromboelastometry
Time Frame: Pre-treatment baseline
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Ticagrelor + ASA + Bivalirudin | Clopidogrel + ASA + Bivalirudin
Number analyzed (Participants) | 15 | 15
seconds | 53.1 [48.8 to 57.5] | 51.1 [45.0 to 57.2]

7. Secondary Outcome: Blood Thrombogenicity
Description: Coagulation times, assessed using the ROTEM thromboelastometry
Time Frame: 1 hr post-treatment
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Ticagrelor + ASA + Bivalirudin | Clopidogrel + ASA + Bivalirudin
Number analyzed (Participants) | 15 | 15
seconds | 163.1 [145.8 to 180.5] | 174.0 [155.5 to 192.5]

8. Secondary Outcome: Blood Thrombogenicity
Description: Coagulation times, assessed using the ROTEM thromboelastometry
Time Frame: 24-hours post-treatment
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Ticagrelor + ASA + Bivalirudin | Clopidogrel + ASA + Bivalirudin
Number analyzed (Participants) | 15 | 15
seconds | 56.1 [50.8 to 61.4] | 54.3 [49.6 to 59.1]

ADVERSE EVENTS:
Time Frame: there were no adverse events
Groups:
- Ticagrelor, Then Clopidogrel; Clopidogrel, Then Ticagrelor: Acute antithrombotic effects of ticagrelor (180 mg + 90 mg) versus clopidogrel (600mg), when coadministered with aspirin (81mg) and bivalirudin (weight-adjusted clinical dose, given as bolus plus 1-hour infusion) with a 1-2 week wash out period in between.
Arm/Group | Ticagrelor, Then Clopidogrel | Clopidogrel, Then Ticagrelor
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes